CLINICAL TRIAL: NCT01522391
Title: A Randomized, Double-blinded Placebo-controlled Study to Investigate Antimicrobial Efficacy and Safety Following Topical Application of DPK-060
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: DermaGen AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DCS-001; 2007-007103-32 (EudraCT Number)
Record Dates: First submitted 2012-01-20; First posted 2012-01-31 (Estimated); Results first posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Ointments

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo for DPK-060 ointment (Placebo Comparator)
  Interventions: Drug: Placebo for DPK-060 ointment
- DPK-060 1% ointment (Experimental)
  Interventions: Drug: DPK-060 1% ointment

INTERVENTIONS:
Drug: DPK-060 1% ointment — DPK-060 1% ointment applied to the skin, two applications per day using approximately 3 mg ointment per cm2
  Arms: DPK-060 1% ointment
Drug: Placebo for DPK-060 ointment — Placebo for DPK-060 ointment applied to the skin, two applications per day using approximately 3 mg ointment per cm2
  Arms: Placebo for DPK-060 ointment

SUMMARY:
The primary objective of this study was to evaluate microbial density in eczematous lesions during two weeks of twice daily therapy with the investigational product, DPK-060 1% ointment, compared with placebo in patients with atopic dermatitis. This randomized, double-blind, placebo-controlled part of the study was preceded with an open-label investigation in a small group of patients (n=5) treated with two applications of DPK-060 1% ointment per day for four days to assess safety, local tolerability and systemic absorption of DPK-060.

The secondary objectives were to evaluate severity of eczema and pruritus, to assess the tolerability and safety of the treatment and to assess the degree of systemic absorption of DPK-060 in blood on Day 7 and Day 21 in a sub-set of 10 patients.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of atopic dermatitis
* Treatable eczematous lesions of a total area of at least 25 cm2 (100 cm2 for the initial five patients)
* Female patients of childbearing potential had to be using an appropriate method of contraception.
* Female patients of childbearing potential were not eligible before PK data from the first 10 patients had been evaluated and the Medical Products Agency (Swedish regulatory agency) had given approval to include women of childbearing potential.

Exclusion Criteria:

* Significant clinical illness, within the two weeks prior to first dose, which could affect the outcome of the study
* Previous local or systemic antimicrobial therapy within the last four weeks prior to the first application of the investigational product (DPK-060 1% or placebo ointment)
* Existence of any surgical or medical condition which, in the judgment of the investigator, might interfere with the absorption, distribution, metabolism or excretion of the drug
* Patients who had had systemic treatment for atopic dermatitis or other topical or transdermal treatments (such as nicotine, hormone replacement therapies)on the site of eczema within 14 days prior to first application of DPK-060 1% or placebo ointment and/or topical treatment with tar, any corticosteroid,topical immunomodulators or oral treatment with any corticosteroids within 14 days prior to first application and/or oral antihistamines within 14 days of the first dose.
* A need for any other medication during the period 0 to 7 days before entry to the study, (excluding the oral contraceptive pill for females) except those deemed by the principal investigator / clinical investigator not to interfere with the outcome of the study
* Diagnosis of other skin diseases, which in the opinion of the investigator, were likely to adversely affect the outcome of the study
* History or evidence of significant cardiac, renal, hepatic or endocrine disease
* Significant hypersensitivity or allergy, as judged by the investigator
* Immunocompromised patients
* Lice or scabies
* Tinea corporis
* Hypersensitivity to the ingredients of the vehicle
* The presence of prominent tattoos at sites of application of DPK-060 1% or placebo ointment
* Donation of blood, exceeding 450 mL, during the three months prior to first dose
* Participation in a clinical study during the 12 weeks prior to first dose
* Ongoing alcohol or drug abuse
* Positive pregnancy test or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Quintiles Hermelinen AB, Luleå, Sweden

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Started | 20 | 21
Completed | 19 | 20
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 21 | 41
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (14.6) | 33.1 (13.5) | 32.5 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  Sweden | 20 | 21 | 41

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Total Microbial Colony Forming Units (CFU) Count at Day 14 Full Analysis Set
Description: The total microbial colony forming units count is the number of CFU/cm2 for total microbial count in eczematous lesions.
Time Frame: Baseline and Day 14
Population: The full analysis set is defined as the patients who received at least one dose of the investigational product and produced study data beyond baseline.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 20 | 21
Percent change | -94 [-100 to 19483] | -100 [-100 to 40926]
Statistical Analysis 1: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Test type: Other; p = 0.012, Mixed Models Analysis; Ratio between geometric means = 0.045, 95% CI 2-sided [0.004 to 0.491]

2. Primary Outcome: Percent Change From Baseline in Total Microbial Colony Forming Units (CFU) Count at Day 14 Per Protocol Analysis Set
Description: The total microbial colony forming units count is the number of CFU/cm2 for total microbial count in eczematous lesions.
Time Frame: Baseline and Day 14
Population: Per protocol analysis set is defined as the patients who completed the study according to the protocol.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 19 | 20
Percent change | -90 [-100 to 19483] | -100 [-100 to -52]
Statistical Analysis 1: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Test type: Other; p = 0.012, Mixed Models Analysis; Ratio between geometric means = 0.045, 95% CI 2-sided [0.004 to 0.491]

3. Secondary Outcome: Percent Change From Baseline in Total Microbial Colony Forming Units (CFU) Count at Day 7 and 21 Full Analysis Set
Description: The total microbial colony forming units count is the number of CFU/cm2 for total microbial count in eczematous lesions.
Time Frame: Baseline, Day 7 and 21
Population: as for outcome 1
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 20 | 21
Percent change
  Day 7 | -73 [-100 to 73429] | -98 [-100 to 40926]
  Day 21 | 14 [-99 to 294067] | -37 [-100 to 40926]
Statistical Analysis 1: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 7; Test type: Other; p = 0.242, Mixed Models Analysis; Ratio between geometric means = 0.242, 95% CI 2-sided [0.022 to 2.66]
Statistical Analysis 2: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 21; Test type: Other; p = 0.482, Mixed Models Analysis; Ratio between geometric means = 0.428, 95% CI 2-sided [0.039 to 4.696]

4. Secondary Outcome: Percent Change From Baseline in Total Microbial Colony Forming Units (CFU) Count at Day 7 and 21 Per Protocol Analysis Set
Description: The total microbial colony forming units count is the number of CFU/cm2 for total microbial count in eczematous lesions.
Time Frame: Baseline, Day 7 and 21
Population: The per protocol analysis set is defined as the patients who completed the study according to the protocol.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 19 | 20
Percent change
  Day 7 | -73 [-100 to 73429] | -96 [-100 to 563]
  Day 21 | 20 [-99 to 294067] | -49 [-100 to 14344]
Statistical Analysis 1: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 7; Test type: Other; p = 0.242, Mixed Models Analysis; Ratio between geometric means = 0.242, 95% CI 2-sided [0.022 to 2.660]
Statistical Analysis 2: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 21; Test type: Other; p = 0.482, Mixed Models Analysis; Ratio between geometric means = 0.428, 95% CI 2-sided [0.039 to 4.696]

5. Secondary Outcome: Percent Change From Baseline in S.Aureus CFU Count at Day 7, 14 and 21 Full Analysis Set
Description: The S.Aureus CFU count is the number of CFU/cm2 for S.Aureus count in eczematous lesions.
Time Frame: Baseline, Day 7, Day 14 and Day 21
Population: as for outcome 1
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 20 | 21
Percent change
  Day 7 | -50 [-100 to 73429] | -100 [-100 to 799900]
  Day 14 | -91 [-100 to 1665] | -100 [-100 to 799900]
  Day 21 | 24 [-100 to 21900] | -2 [-100 to 799900]
Statistical Analysis 1: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 7; Test type: Other; p = 0.395, Mixed Models Analysis; Ratio between geometric means = 0.288, 95% CI 2-sided [0.016 to 5.221]
Statistical Analysis 2: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 14; Test type: Other; p = 0.067, Mixed Models Analysis; Ratio between geometric means = 0.067, 95% CI 2-sided [0.004 to 1.218]
Statistical Analysis 3: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 21; Test type: Other; p = 0.620, Mixed Models Analysis; Ratio between geometric means = 0.484, 95% CI 2-sided [0.027 to 8.787]

6. Secondary Outcome: Percent Change From Baseline in S.Aureus CFU Count at Day 7, 14 and 21 Per Protocol Analysis Set
Description: The S.Aureus CFU count is the number of CFU/cm2 for S.Aureus count in eczematous lesions.
Time Frame: Baseline, Day 7, Day 14 and Day 21
Population: The per protocol analysis set is defined as the patients who completed the study according to the protocol.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 19 | 20
Percent change
  Day 7 | -60 [-100 to 73429] | -100 [-100 to 546]
  Day 14 | -91 [-100 to 1665] | -100 [-100 to -77]
  Day 21 | 24 [-100 to 21900] | -36 [-100 to 3614]
Statistical Analysis 1: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 7; Test type: Other; p = 0.403, Mixed Models Analysis; Ratio between geometric means = 0.287, 95% CI 2-sided [0.015 to 5.550]
Statistical Analysis 2: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 14; Test type: Other; p = 0.021, Mixed Models Analysis; Ratio between geometric means = 0.032, 95% CI 2-sided [0.002 to 0.583]
Statistical Analysis 3: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 21; Test type: Other; p = 0.368, Mixed Models Analysis; Ratio between geometric means = 0.271, 95% CI 2-sided [0.015 to 4.779]

7. Secondary Outcome: Percent Change From Baseline in KNS CFU Count at Day 7, 14 and 21 Full Analysis Set
Description: The KNS CFU count is the number of CFU/cm2 for coagulase-negative staphylococcus count in eczematous lesions.
Time Frame: Baseline, Day 7, Day 14 and Day 21
Population: as for outcome 1
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 20 | 21
Percent change
  Day 7 | -99 [-100 to 93] | -100 [-100 to 353]
  Day 14 | -95 [-100 to 233] | -100 [-100 to -52]
  Day 21 | -82 [-100 to 1694] | -78 [-100 to 6844]
Statistical Analysis 1: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 7; Test type: Other; p = 0.970, Mixed Models Analysis; Ratio between geometric means = 1.045, 95% CI 2-sided [0.106 to 10.32]
Statistical Analysis 2: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 14; Test type: Other; p = 0.009, Mixed Models Analysis; Ratio between geometric means = 0.045, 95% CI 2-sided [0.005 to 0.447]
Statistical Analysis 3: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 21; Test type: Other; p = 0.377, Mixed Models Analysis; Ratio between geometric means = 0.360, 95% CI 2-sided [0.036 to 3.556]

8. Secondary Outcome: Percent Change From Baseline in KNS CFU Count at Day 7, 14 and 21 Per Protocol Analysis Set
Description: The KNS CFU count is the number of CFU/cm2 for coagulase-negative staphylococcus count in eczematous lesions.
Time Frame: Baseline, Day 7, Day 14 and Day 21
Population: The per protocol analysis set is defined as the patients who completed the study according to the protocol.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 19 | 20
Percent change
  Day 7 | -99 [-100 to 93] | -98 [-100 to 353]
  Day 14 | -93 [-100 to 233] | -100 [-100 to -52]
  Day 21 | -82 [-100 to 1694] | -73 [-100 to 6844]
Statistical Analysis 1: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 7; Test type: Other; p = 0.974, Mixed Models Analysis; Ratio between geometric means = 0.961, 95% CI 2-sided [0.081 to 11.43]
Statistical Analysis 2: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 14; Test type: Other; p = 0.013, Mixed Models Analysis; Ratio between geometric means = 0.046, 95% CI 2-sided [0.004 to 0.512]
Statistical Analysis 3: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 21; Test type: Other; p = 0.504, Mixed Models Analysis; Ratio between geometric means = 0.447, 95% CI 2-sided [0.041 to 4.883]

9. Secondary Outcome: Percent Change From Baseline in Gram-positive Bacteria CFU Count at Day 7, 14 and 21 Full Analysis Set
Description: The gram-positive CFU count is the number of CFU/cm2 for gram-positive bacteria count in eczematous lesions.
Time Frame: Baseline, Day 7, Day 14 and Day 21
Population: as for outcome 1
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 20 | 21
Percent change
  Day 7 | -73 [-100 to 73429] | -98 [-100 to 40926]
  Day 14 | -94 [-100 to 19483] | -100 [-100 to 40926]
  Day 21 | 14 [-99 to 291567] | -37 [-100 to 40926]
Statistical Analysis 1: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 7; Test type: Other; p = 0.242, Mixed Models Analysis; Ratio between geometric means = 0.242, 95% CI 2-sided [0.022 to 2.659]
Statistical Analysis 2: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 14; Test type: Other; p = 0.012, Mixed Models Analysis; Ratio between geometric means = 0.045, 95% CI 2-sided [0.004 to 0.491]
Statistical Analysis 3: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 21; Test type: Other; p = 0.483, Mixed Models Analysis; Ratio between geometric means = 0.428, 95% CI 2-sided [0.039 to 4.697]

10. Secondary Outcome: Percent Change From Baseline in Gram-positive Bacteria CFU Count at Day 7, 14 and 21 Per Protocol Analysis Set
Description: The gram-positive bacteria CFU count is the number of CFU/cm2 for gram-positive bacteria count in eczematous lesions.
Time Frame: Baseline, Day 7, Day 14 and Day 21
Population: The per protocol analysis set is defined as the patients who completed the study according to the protocol.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 19 | 20
Percent change
  Day 7 | -73 [-100 to 73429] | -96 [-100 to 563]
  Day 14 | -90 [-100 to 19483] | -100 [-100 to -52]
  Day 21 | 20 [-99 to 291567] | -49 [-100 to 14344]
Statistical Analysis 1: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 7; Test type: Other; p = 0.197, Mixed Models Analysis; Ratio between geometric means = 0.202, 95% CI 2-sided [0.017 to 2.340]
Statistical Analysis 2: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 14; Test type: Other; p = 0.002, Mixed Models Analysis; Ratio between geometric means = 0.021, 95% CI 2-sided [0.002 to 0.227]
Statistical Analysis 3: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 21; Test type: Other; p = 0.257, Mixed Models Analysis; Ratio between geometric means = 0.257, 95% CI 2-sided [0.024 to 2.752]

11. Secondary Outcome: Change in Total Treated Eczema Area Full Analysis Set
Description: Change from baseline (Day 1 morning) in total treated eczema area measured in cm2.
Time Frame: Baseline, Day 7, Day 14 and Day 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 20 | 21
cm2
  Day 7 | 12.0 (32.8) | 32.3 (92.2)
  Day 14 | -15.0 (42.9) | 14.1 (82.7)
  Day 21 | 17.4 (78.7) | 5.8 (60.8)
Statistical Analysis 1: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 7; Test type: Other; p = 0.346, Mixed Models Analysis; Least Square Mean Difference = 20.38, 95% CI 2-sided [-22.42 to 63.19]
Statistical Analysis 2: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 14; Test type: Other; p = 0.18, Mixed Models Analysis; Least Square Mean Difference = 29.10, 95% CI 2-sided [-13.71 to 71.90]
Statistical Analysis 3: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 21; Test type: Other; p = 0.590, Mixed Models Analysis; Least Square Mean Difference = -11.64, 95% CI 2-sided [-54.44 to 31.16]

12. Secondary Outcome: Change in Total Treated Eczema Area Per Protocol Analysis Set
Description: Change from baseline (Day 1 morning) in total treated eczema area measured in cm2.
Time Frame: Baseline, Day 7, Day 14 and Day 21
Population: The per protocol analysis set is defined as the patients who completed the study according to the protocol.
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 19 | 20
cm2
  Day 7 | 12.1 (33.7) | 18.0 (66.4)
  Day 14 | -16.0 (44.9) | -1.2 (45.4)
  Day 21 | 21.1 (82.4) | 2.4 (60.3)
Statistical Analysis 1: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 7; Test type: Other; p = 0.748, Mixed Models Analysis; Least Square Mean Difference = 5.95, 95% CI 2-sided [-30.84 to 42.73]
Statistical Analysis 2: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 14; Test type: Other; p = 0.437, Mixed Models Analysis; Least Square Mean Difference = 14.62, 95% CI 2-sided [-22.65 to 51.88]
Statistical Analysis 3: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 21; Test type: Other; p = 0.322, Mixed Models Analysis; Least Square Mean Difference = -18.66, 95% CI 2-sided [-55.92 to 18.61]

13. Secondary Outcome: Change in Area of Microbial Counting Site Full Analysis Set
Description: Change from baseline (Day 1 morning) in area of microbial counting site measured in cm2.
Time Frame: Baseline, Day 7, Day 14 and Day 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 20 | 21
cm2
  Day 7 | 12.1 (25.5) | 20.1 (68.0)
  Day 14 | -16.3 (32.2) | 4.2 (49.1)
  Day 21 | 8.9 (66.0) | 7.6 (62.3)
Statistical Analysis 1: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 7; Test type: Other; p = 0.631, Mixed Models Analysis; Least Square Mean Difference = 8.04, 95% CI 2-sided [-25.15 to 41.24]
Statistical Analysis 2: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 14; Test type: Other; p = 0.224, Mixed Models Analysis; Least Square Mean Difference = 20.44, 95% CI 2-sided [-12.75 to 53.63]
Statistical Analysis 3: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 21; Test type: Other; p = 0.941, Mixed Models Analysis; Least Square Mean Difference = -1.23, 95% CI 2-sided [-34.42 to 31.96]

14. Secondary Outcome: Change in Area of Microbial Counting Site Per Protocol Analysis Set
Description: Change from baseline (Day 1 morning) in area of microbial counting site measured in cm2.
Time Frame: Baseline, Day 7, Day 14 and Day 21
Population: The per protocol analysis set is defined as the patients who completed the study according to the protocol.
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 19 | 20
cm2
  Day 7 | 13.3 (26.7) | 15.3 (66.0)
  Day 14 | -18.2 (33.4) | -1.5 (42.8)
  Day 21 | 9.8 (69.7) | 2.2 (58.5)
Statistical Analysis 1: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 7; Test type: Other; p = 0.954, Mixed Models Analysis; Least Square Means Difference = 0.97, 95% CI 2-sided [-32.93 to 34.87]
Statistical Analysis 2: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 14; Test type: Other; p = 0.358, Mixed Models Analysis; Least Square Mean Difference = 15.72, 95% CI 2-sided [-18.18 to 49.62]
Statistical Analysis 3: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 21; Test type: Other; p = 0.642, Mixed Models Analysis; least Square Mean Difference = -7.94, 95% CI 2-sided [-41.82 to 25.94]

15. Secondary Outcome: Erythema Eczema Area and Severity Index (EASI) Full Analysis Set
Description: Evaluation of erythema on a scale 0-3 where 0=No symptoms, 1=Slight, 2=Moderate, 3=Severe
Time Frame: Day 7, Day 14 and Day 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 20 | 21
Participants
  Day 7: No symptoms | 0 | 0
  Day 7: Slight | 11 | 13
  Day 7: Moderate | 8 | 7
  Day 7: Severe | 1 | 1
  Day 14: No symptoms | 0 | 0
  Day 14: Slight | 11 | 11
  Day 14: Moderate | 8 | 9
  Day 14: Severe | 1 | 1
  Day 21: No symptoms | 0 | 0
  Day 21: Slight | 10 | 14
  Day 21: Moderate | 8 | 6
  Day 21: Severe | 2 | 1
Statistical Analysis 1: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 7; Test type: Other; p = 0.701, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 14; Test type: Other; p = 0.898, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 21; Test type: Other; p = 0.271, Cochran-Mantel-Haenszel

16. Secondary Outcome: Erythema Eczema Area and Severity Index (EASI) Per Protocol Analysis Set
Description: Evaluation of erythema on a scale 0-3 where 0=No symptoms, 1=Slight, 2=Moderate, 3=Severe
Time Frame: Day 7, Day 14 and Day 21
Population: The per protocol analysis set is defined as the patients who completed the study according to the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 19 | 20
Participants
  Day 7: No symptoms | 0 | 0
  Day 7: Slight | 10 | 13
  Day 7: Moderate | 8 | 6
  Day 7: Severe | 1 | 1
  Day 7: Missing | 0 | 0
  Day 14: No symptoms | 0 | 0
  Day 14: Slight | 9 | 11
  Day 14: Moderate | 8 | 8
  Day 14: Severe | 1 | 1
  Day 14: Missing | 1 | 0
  Day 21: No symptoms | 0 | 0
  Day 21: Slight | 8 | 13
  Day 21: Moderate | 8 | 6
  Day 21: Severe | 2 | 1
  Day 21: Missing | 1 | 0
Statistical Analysis 1: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 7; Test type: Other; p = 0.511, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 14; Test type: Other; p = 0.777, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 21; Test type: Other; p = 0.204, Cochran-Mantel-Haenszel

17. Secondary Outcome: Excoriations Eczema Area and Severity Index (EASI) Full Analysis Set
Description: Evaluation of excoriations on a scale 0-3 where 0=No symptoms, 1=Slight, 2=Moderate, 3=Severe
Time Frame: Day 7, Day 14 and Day 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 20 | 21
Participants
  Day 7: No symptoms | 5 | 6
  Day 7: Slight | 7 | 10
  Day 7: Moderate | 6 | 3
  Day 7: Severe | 2 | 2
  Day 14: No symptoms | 6 | 9
  Day 14: Slight | 7 | 8
  Day 14: Moderate | 7 | 4
  Day 14: Severe | 0 | 0
  Day 21: No symptoms | 5 | 8
  Day 21: Slight | 6 | 9
  Day 21: Moderate | 8 | 4
  Day 21: Severe | 1 | 0
Statistical Analysis 1: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 7; Test type: Other; p = 0.489, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 14; Test type: Other; p = 0.249, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 21; Test type: Other; p = 0.098, Cochran-Mantel-Haenszel

18. Secondary Outcome: Excoriations Eczema Area and Severity Index (EASI) Per Protocol Analysis Set
Description: Evaluation of excoriations on a scale 0-3 where 0=No symptoms, 1=Slight, 2=Moderate, 3=Severe
Time Frame: Day 7, Day 14 and Day 21
Population: The per protocol analysis set is defined as the patients who completed the study according to the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 19 | 20
Participants
  Day 7: No symptoms | 4 | 6
  Day 7: Slight | 7 | 10
  Day 7: Moderate | 6 | 2
  Day 7: Severe | 2 | 2
  Day 7: Missing | 0 | 0
  Day 14: No symptoms | 5 | 9
  Day 14: Slight | 6 | 8
  Day 14: Moderate | 7 | 3
  Day 14: Severe | 0 | 0
  Day 14: Missing | 1 | 0
  Day 21: No symptoms | 3 | 8
  Day 21: Slight | 6 | 8
  Day 21: Moderate | 8 | 4
  Day 21: Severe | 1 | 0
  Day 21: Missing | 1 | 0
Statistical Analysis 1: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 7; Test type: Other; p = 0.291, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: DPK-060 1% Ointment; Day 14; Test type: Other; p = 0.113, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 21; Test type: Other; p = 0.033, Cochran-Mantel-Haenszel

19. Secondary Outcome: Infiltration Eczema Area and Severity Index (EASI) Full Analysis Set
Description: Evaluation of infiltration on a scale 0-3 where 0=No symptoms, 1=Slight, 2=Moderate, 3=Severe
Time Frame: Day 7, Day 14 and Day 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 20 | 21
Participants
  Day 7: No symptoms | 4 | 4
  Day 7: Slight | 13 | 12
  Day 7: Moderate | 2 | 5
  Day 7: Severe | 1 | 0
  Day 14: No symptoms | 5 | 5
  Day 14: Slight | 9 | 11
  Day 14: Moderate | 6 | 5
  Day 14: Severe | 0 | 0
  Day 21: No symptoms | 5 | 7
  Day 21: Slight | 7 | 9
  Day 21: Moderate | 6 | 5
  Day 21: Severe | 2 | 0
Statistical Analysis 1: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 7; Test type: Other; p = 0.825, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 14; Test type: Other; p = 0.825, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Test type: Other; p = 0.208, Cochran-Mantel-Haenszel

20. Secondary Outcome: Infiltration Eczema Area and Severity Index (EASI) Per Protocol Analysis Set
Description: Evaluation of infiltration on a scale 0-3 where 0=No symptoms, 1=Slight, 2=Moderate, 3=Severe
Time Frame: Day 7, Day 14 and Day 21
Population: The per protocol analysis set is defined as the patients who completed the study according to the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 19 | 20
Participants
  Day 7: No symptoms | 4 | 4
  Day 7: Slight | 12 | 11
  Day 7: Moderate | 2 | 5
  Day 7: Severe | 1 | 0
  Day 7: Missing | 0 | 0
  Day 14: No symptoms | 5 | 5
  Day 14: Slight | 7 | 10
  Day 14: Moderate | 6 | 5
  Day 14: Severe | 0 | 0
  Day 14: Missing | 1 | 0
  Day 21: No symptoms | 3 | 7
  Day 21: Slight | 7 | 8
  Day 21: Moderate | 6 | 5
  Day 21: Severe | 2 | 0
  Day 21: Missing | 1 | 0
Statistical Analysis 1: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 7; Test type: Other; p = 0.825, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 14; Test type: Other; p = 0.820, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 21; Test type: Other; p = 0.086, Cochran-Mantel-Haenszel

21. Secondary Outcome: Lichenification Eczema Area and Severity Index (EASI) Full Analysis Set
Description: Evaluation of lichenification on a scale 0-3 where 0=No symptoms, 1=Slight, 2=Moderate, 3=Severe
Time Frame: Day 7, Day 14 and Day 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 20 | 21
Participants
  Day 7: No symptoms | 0 | 3
  Day 7: Slight | 14 | 12
  Day 7: Moderate | 6 | 6
  Day 7: Severe | 0 | 0
  Day 14: No symptoms | 4 | 4
  Day 14: Slight | 9 | 10
  Day 14: Moderate | 7 | 7
  Day 14: Severe | 0 | 0
  Day 21: No symptoms | 4 | 1
  Day 21: Slight | 8 | 15
  Day 21: Moderate | 8 | 5
  Day 21: Severe | 0 | 0
Statistical Analysis 1: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 7; Test type: Other; p = 0.378, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 14; Test type: Other; p = 0.975, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 21; Test type: Other; p = 0.962, Cochran-Mantel-Haenszel

22. Secondary Outcome: Lichenification Eczema Area and Severity Index (EASI) Per Protocol Analysis Set
Description: Evaluation of lichenification on a scale 0-3 where 0=No symptoms, 1=Slight, 2=Moderate, 3=Severe
Time Frame: Day 7, Day 14 and Day 21
Population: The per protocol analysis set is defined as the patients who completed the study according to the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 19 | 20
Participants
  Day 7: No symptoms | 0 | 3
  Day 7: Slight | 13 | 11
  Day 7: Moderate | 6 | 6
  Day 7: Severe | 0 | 0
  Day 7: Missing | 0 | 0
  Day 14: No symptoms | 4 | 4
  Day 14: Slight | 7 | 9
  Day 14: Moderate | 7 | 7
  Day 14: Severe | 0 | 0
  Day 14: Missing | 1 | 0
  Day 21: No symptoms | 2 | 1
  Day 21: Slight | 8 | 14
  Day 21: Moderate | 8 | 5
  Day 21: Severe | 0 | 0
  Day 21: Missing | 1 | 0
Statistical Analysis 1: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 7; Test type: Other; p = 0.375, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 14; Test type: Other; p = 0.946, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 21; Test type: Other; p = 0.495, Cochran-Mantel-Haenszel

23. Secondary Outcome: Investigator's Global Assessment of Eczema Change Full Analysis Set
Description: Investigator's global assessment of eczema status since previous dose application on a categorical scale (worse, unchanged, improved)
Time Frame: Day 7, Day 14 and Day 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 20 | 21
Participants
  Day 7: Worse | 4 | 4
  Day 7: Unchanged | 8 | 6
  Day 7: Improved | 8 | 11
  Day 14: Worse | 5 | 3
  Day 14: Unchanged | 4 | 9
  Day 14: Improved | 11 | 9
  Day 21: Worse | 10 | 5
  Day 21: Unchanged | 6 | 10
  Day 21: Improved | 4 | 6

24. Secondary Outcome: Investigator's Global Assessment of Eczema Change Per Protocol Analysis Set
Description: as for outcome 23
Time Frame: Day 7, Day 14 and Day 21
Population: The per protocol analysis set is defined as the patients who completed the study according to the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 19 | 20
Participants
  Day 7: Worse | 4 | 3
  Day 7: Unchanged | 7 | 6
  Day 7: Improved | 8 | 11
  Day 7: Missing | 0 | 0
  Day 14: Worse | 5 | 2
  Day 14: Unchanged | 3 | 9
  Day 14: Improved | 10 | 9
  Day 14: Missing | 1 | 0
  Day 21: Worse | 10 | 5
  Day 21: Unchanged | 6 | 9
  Day 21: Improved | 2 | 6
  Day 21: Missing | 1 | 0

25. Secondary Outcome: Change From Baseline in Visual Analog Scale of Itching (VASI) Full Analysis Set
Description: The Visual Analog Scale of Itching (VASI), is the patient's assessment of itching on a 0-100 mm scale. 0 mm corresponds to no itching and 100 mm corresponds to maximum itching. Change from baseline is the change from day 1 morning.
Time Frame: Baseline, Day 7, Day 14 and Day 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 20 | 21
mm
  Day 7 | -11.19 (26.19) | -15.19 (27.23)
  Day 14 | -15.34 (21.28) | -10.60 (25.97)
  Day 21 | -4.34 (28.66) | -13.41 (27.72)
Statistical Analysis 1: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 7 morning; Test type: Other; p = 0.477, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 14 morning; Test type: Other; p = 0.651, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 21 morning; Test type: Other; p = 0.340, Wilcoxon (Mann-Whitney)

26. Secondary Outcome: Change From Baseline in Visual Analog Scale of Itching (VASI) Per Protocol Analysis Set
Description: as for outcome 25
Time Frame: Baseline, Day 7, Day 14 and Day 21
Population: The per protocol analysis set is defined as the patients who completed the study according to the protocol.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 19 | 20
mm
  Day 7 | -11.32 (26.90) | -20.48 (18.72)
  Day 14 | -16.91 (24.25) | -14.92 (18.37)
  Day 21 | -2.24 (29.44) | -12.89 (28.34)
Statistical Analysis 1: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 7 morning; Test type: Other; p = 0.300, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 14; Test type: Other; p = 0.705, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo for DPK-060 Ointment vs DPK-060 1% Ointment; Day 21; Test type: Other; p = 0.286, Wilcoxon (Mann-Whitney)

27. Secondary Outcome: Patient's Global Assessment of Eczema Change Full Analysis Set
Description: Patient's global assessment of eczema status since previous dose application on a categorical scale (worse, unchanged, improved)
Time Frame: Day 7, Day 14 and Day 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 20 | 21
Participants
  Day 7: Worse | 1 | 2
  Day 7: Unchanged | 14 | 14
  Day 7: Improved | 5 | 5
  Day 14 morning: Worse | 0 | 2
  Day 14 morning: Unchanged | 13 | 13
  Day 14 morning: Improved | 7 | 6
  Day 21: Worse | 7 | 5
  Day 21: Unchanged | 9 | 8
  Day 21: Improved | 4 | 8

28. Secondary Outcome: Patient's Global Assessment of Eczema Change Per Protocol Analysis Set
Description: as for outcome 27
Time Frame: Day 7, Day 14 and Day 21
Population: The per protocol analysis set is defined as the patients who completed the study according to the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Number analyzed (Participants) | 19 | 20
Participants
  Day 7: Worse | 1 | 0
  Day 7: Unchanged | 14 | 13
  Day 7: Improved | 4 | 5
  Day 7: Missing | 0 | 2
  Day 14 morning: Worse | 0 | 1
  Day 14 morning: Unchanged | 9 | 12
  Day 14 morning: Improved | 5 | 5
  Day 14 morning: Missing | 5 | 2
  Day 21: Worse | 7 | 5
  Day 21: Unchanged | 8 | 8
  Day 21: Improved | 2 | 7
  Day 21: Missing | 2 | 0

ADVERSE EVENTS:
Arm/Group | Placebo for DPK-060 Ointment | DPK-060 1% Ointment
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 7/20 | 10/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo for DPK-060 Ointment (N=20) | DPK-060 1% Ointment (N=21)
Nasopharyngitis (Infections and infestations) | 0 | 3
Headache (Nervous system disorders) | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 4
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes